CLINICAL TRIAL: NCT01027208
Title: A Rollover Study of Ixabepilone (BMS-247550) In Patients With Metastatic Breast Cancer Previously Treated With An Anthracycline And Who Are Taxane Resistant Who Have Completed Study CA163107 And Who Are Benefiting From Continuation On Therapy With Ixabepilone
Brief Title: A Rollover Study of Ixabepilone (BMS-247550) In Patients With Metastatic Breast Cancer Previously Treated With An Anthracycline
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-130
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixabepilone (Experimental)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Lyophilized and solvent, IV, 10-50 mg/m²
  Other Names: Ixempra

SUMMARY:
To provide extended access to Ixabepilone therapy to subjects with metastatic breast cancer who have completed the previous Phase II study (CA163-107)

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 years or older
* Patients with metastatic breast cancer whose primary lesion was definitely diagnosed to be breast by histological or cellular examination

Exclusion Criteria:

* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≥2

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Provide extended access to Ixabepilone therapy to subjects with metastatic breast cancer who have completed the previous Phase II study (CA163107) and are benefiting from continuation on therapy with Ixabepilone as determined by the treating investigator | 21-day cycles until documented disease progression or unacceptable toxicity
To evaluate the frequency and the severity of observed adverse reactions in treated patients, graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 | 21-day cycles until documented disease progression or unacceptable toxicity

SECONDARY OUTCOMES:
Secondary objectives will be assessed by combining data with the previous Phase II study CA163107 | 21-day cycles until documented disease progression or unacceptable toxicity
To evaluate the antitumor response according to the RECIST criteria | 21-day cycles until documented disease progression or unacceptable toxicity
To evaluate the duration of achieved responses | 21-day cycles until documented disease progression or unacceptable toxicity
To evaluate time to progression (TTP) | 21-day cycles until documented disease progression or unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- Japan (14):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kashiwa-Shi, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Matabashi-Shi, Gunma
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Isehara-Shi, Kanagawa
  - Local Institution, Niigata, Niigata
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Saitama, Saitama
  - Local Institution, Utsunomiya, Tochigi
  - Local Institution, Bunkyo-Ku, Tokyo
  - Local Institution, Chuo-Ku, Tokyo
  - Local Institution, Tokyo, Tokyo
  - Local Institution, Toshima-Ku, Tokyo

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx